CLINICAL TRIAL: NCT06945809
Title: Guo&Amp;'s Distal Entry Tear Repair: a Multicenter, Prospective, Superiority, Randomized Controlled Trial of the Novel WeFlow-EndoPatch Aortic Endovascular Patch System
Brief Title: Guo&Amp;'s Distal Entry Tear Repair With WeFlow-EndoPatch System (Gallant Study)
Acronym: Gallant
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WQ11-2402
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Aortic Dissection; Distal Entry Tear
Keywords: Aortic Dissection; Distal tear; descending aorta
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EndoPatch Group (Experimental): Subject in this group will receive treatment with the WeFlow-EndoPatch Aortic Endovascular Patch System.
  Interventions: Device: WeFlow-EndoPatch Aortic Endovascular Patch System
- Control Group (Other): Subject in this group will receive conventional treatment.
  Interventions: Other: Conventional Treatment group

INTERVENTIONS:
Device: WeFlow-EndoPatch Aortic Endovascular Patch System — The WeFlow-EndoPatch Aortic Endovascular Patch System for aortic dissection tear is composed of a dissection tear patch system and an adjustable bend conveyor. The patch system is composed of a patch and a conveying steel cable. The patch is pre-installed on the conveying steel cable.
  Arms: EndoPatch Group
Other: Conventional Treatment group — Doctors prescribe conventional medicines and regular imaging tests.
  Arms: Control Group

SUMMARY:
A Multicenter, Randomized Controlled Study About the Safety and Efficacy of WeFlow-EndoPatch Aortic Endovascular Patch System manufactured by EndoNom Medtech (Hangzhou) Co., Ltd. for Chronic Aortic Dissection . (GALLANT Study)

DETAILED DESCRIPTION:
This study is a multicenter, prospective, superiority, randomized controlled trial about the safety and efficacy of WeFlow-EndoPatch Aortic Endovascular Patch System. It is expected to complete the implantation of 204 patients in 15 centers within 24 months, and interim follow-up was conducted before discharge, 30 days after surgery, 6 months after surgery and 12 months after surgery, long-term follow-up will be performed at 24th month, 36th month, 48th month and 60th month postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years old, no gender limitation;
* The patient was diagnosed with chronic aortic dissection after the repair of the main artery dissection, with distal tears required seal;
* The maximum diameter of the descending thoracic aorta is 3.5-5cm；
* The number of thoracic descending aorta tears is ≤2, and the maximum diameter of the tears is 2-30 mm；
* With appropriate artery approaches, endovascular treatment can be performed；
* Those who can understand the purpose of the trial, voluntarily participate in the study, sign the informed consent form by themselves or their legal representative, and are willing to complete the follow-up according to the protocol requirements.

Exclusion Criteria:

* Rupture or threatened rupture of aortic dissection;
* Proximal type I internal leakage after aortic repair;
* New distal SINE;
* Abdominal aortic dissection aneurysm diameter ≥5 cm;
* The edge of the tear from the opening of celiac trunk is<4 mm;
* The same operation requires intervention in other vascular diseases (such as coronary artery, renal artery, superior mesenteric artery, etc.);
* Acute systemic infection;
* History of myocardial infarction, TIA or cerebral infarction within the past 3 months;
* Cardiac function Grade IV (NYHA rating) or LVEF < 30%;
* Hematological abnormalities: leukopenia (WBC < 3×10^9/L), anemia (Hb < 90 g/L); Coagulation dysfunction, thrombocytopenia (PLT count < 50×10^9/L);
* Renal insufficiency: serum creatinine > 150 umol/L (or 3.0 mg/dL) and/or advanced kidney disease requiring renal dialysis, as determined by the investigator after thorough analysis;
* Severe liver insufficiency: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeds the normal upper limit by 5 times; Serum total bilirubin (STB) exceeded the normal upper limit by 2 times;
* Allergic to contrast agents, anesthetics, patchs, and delivery materials;
* Pregnant or breastfeeding;
* Participated in clinical trials of other drugs or devices during the same period;
* Life expectancy is less than 12 months (such as advanced malignant tumors); Investigator judged that not suitable for interventional treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Treatment Success Rate | 12 months
  The success rate of aortic dissection treatment at 12 months is a composite index, including immediate technical success after surgery, freedom from death or aortic dissection rupture, positive aortic remodeling, and freedom from device and/or procedure related reinterventions.

SECONDARY OUTCOMES:
Immediate Technical Success in EndoPatch Group | Immediately after the surgery
  Immediate technical success is defined as successful delivery of the endopatch conveyors to their predetermined positions, accurate positioning and successful deployment of the patch, safe removal of the delivery device outside the body, and no conversion to thoracotomy.
Entry Tears Closure Success in EndoPatch Group | 30 days, 6 months, and 12 months
  Entry tears closure success is defined as absence of TL or FL backflow through the tears on CTA.
False Lumen Thrombosis of the Descending Thoracic Aorta | 30 days, 6 months, and 12 months
  False lumen thrombosis of the descending thoracic aorta (no thrombosis, partial thrombosis, complete thrombosis) observed by postoperative CTA review.
True Lumen/False Lumen/Maximum Total Diameter of Descending Thoracic Aorta | 30 days, 6 months, and 12 months
  True lumen diameter, false lumen diameter and maximum total diameter of the descending thoracic aorta observed by postoperative CTA review.
Device and/or Procedure Related Reinterventions | 30 days, 6 months, and 12 months
No major adverse events within 30 days after surgery | Before discharge, 30 days after surgery
  Major adverse events within 30 days after surgery refer to all-cause death, aortic dissection rupture, myocardial infarction, ischemic stroke, respiratory failure, renal failure, intestinal necrosis, paraplegia, and amputation.
Patch Fall-off in EndoPatch Group | 30 days, 6 months, and 12 months
All-cause Mortality, Aortic Dissection-related Mortality, Serious Adverse Events, and Device-related Adverse Events | 30 days, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Principal Investigator — Chinese PLA Gencral Hosptial

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Erbel R, Aboyans V, Boileau C, Bossone E, Bartolomeo RD, Eggebrecht H, Evangelista A, Falk V, Frank H, Gaemperli O, Grabenwoger M, Haverich A, Iung B, Manolis AJ, Meijboom F, Nienaber CA, Roffi M, Rousseau H, Sechtem U, Sirnes PA, Allmen RS, Vrints CJ; ESC Committee for Practice Guidelines. 2014 ESC Guidelines on the diagnosis and treatment of aortic diseases: Document covering acute and chronic aortic diseases of the thoracic and abdominal aorta of the adult. The Task Force for the Diagnosis and Treatment of Aortic Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2014 Nov 1;35(41):2873-926. doi: 10.1093/eurheartj/ehu281. Epub 2014 Aug 29. No abstract available. PMID 25173340
- [Result] Hofferberth SC, Nixon IK, Mossop PJ. Aortic false lumen thrombosis induction by embolotherapy (AFTER) following endovascular repair of aortic dissection. J Endovasc Ther. 2012 Aug;19(4):538-45. doi: 10.1583/JEVT-12-3844R.1. PMID 22891838
- [Result] Kolbel T, Tsilimparis N, Wipper S, Larena-Avellaneda A, Diener H, Carpenter SW, Debus ES. TEVAR for chronic aortic dissection - is covering the primary entry tear enough? J Cardiovasc Surg (Torino). 2014 Aug;55(4):519-27. Epub 2014 Jun 11. PMID 24918196
- [Result] Zhu C, Huang B, Zhao J, Ma Y, Yuan D, Yang Y, Xiong F, Wang T. Influence of distal entry tears in acute type B aortic dissection after thoracic endovascular aortic repair. J Vasc Surg. 2017 Aug;66(2):375-385. doi: 10.1016/j.jvs.2016.12.142. Epub 2017 Apr 21. PMID 28438361
- [Result] Wojciechowski J, Znaniecki L, Kaszubowski M, Rogowski J. Late Aortic Remodeling after Endovascular Repair of Complicated Type B Aortic Dissection-TEVAR Protects Only the Covered Segment of Thoracic Aorta. Ann Vasc Surg. 2019 Feb;55:148-156. doi: 10.1016/j.avsg.2018.05.057. Epub 2018 Aug 4. PMID 30081168
- [Result] David TE. Adventitial inversion in the distal anastomosis in surgical treatment of acute DeBakey type I aortic dissection. J Thorac Cardiovasc Surg. 2016 May;151(5):1346-7. doi: 10.1016/j.jtcvs.2016.01.028. Epub 2016 Jan 22. No abstract available. PMID 26874601
- [Result] Nienaber CA, Yuan X, Aboukoura M, Blanke P, Jakob R, Janosi RA, Lovato L, Riambau V, Trebacz J, Trimarchi S, Zipfel B, van den Berg JC; ASSIST study group. Improved Remodeling With TEVAR and Distal Bare-Metal Stent in Acute Complicated Type B Dissection. Ann Thorac Surg. 2020 Nov;110(5):1572-1579. doi: 10.1016/j.athoracsur.2020.02.029. Epub 2020 Mar 20. PMID 32205112